CLINICAL TRIAL: NCT00369967
Title: "Quick Start" Initiation of the Contraceptive Vaginal Ring in Adolescents: A Randomized Controlled Trial
Brief Title: Quick Start Initiation of the Contraceptive Vaginal Ring in Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in subject recruitment
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5120008FN
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Contraception Desired
Keywords: Contraception; Adolescents; Contraceptive vaginal ring; Quick start
MeSH Terms: interventions — NuvaRing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quick start (Experimental): Start contraceptive method (NuvaRing) day of enrollment
  Interventions: Drug: NuvaRing
- Traditional start (Active Comparator): Start contraceptive method (NuvaRing) after next menses (per package insert)
  Interventions: Drug: NuvaRing

INTERVENTIONS:
Drug: NuvaRing — Initiation of NuvaRing for contraception
  Other Names: contraceptive vaginal ring

SUMMARY:
We hypothesize that using "quick start" initiation of the contraceptive vaginal ring in adolescents seeking birth control will improve compliance compared to traditional start. We will conduct a randomized controlled trial comparing "quick start" to traditional start initiation of the contraceptive vaginal ring in adolescents seeking birth control. The primary study outcome is method continuation at 3, 6, and 12 months. Secondary outcomes include abnormal bleeding, product satisfaction, and adverse events.

DETAILED DESCRIPTION:
Pregnancy prevention is an important aspect of adolescent healthcare. Adherence to a chosen contraception method is essential to its success. Adolescents are notoriously poor at complying with oral contraceptives (OCs), with continuation rates at one year as low as 12% (1). In those patients who continue their contraceptive method, our best data estimates that the average OC user misses three pills per cycle (2). Given the already highly fluctuant serum hormone levels in OC users (3), this leaves poorly compliant users at greater risk for unintended pregnancy.

The contraceptive vaginal ring is a reliable method of contraception and may be particularly useful in the adolescent population because of its simple monthly dosing schedule (4). It is a combined hormonal contraceptive containing etonogestrel (a progesterone) and ethinyl estradiol (an estrogen), which are released continuously at low levels. The vaginal ring has been shown to have comparable efficacy and tolerability to OCs (5), but does not require daily dosing due to its novel drug delivery system. Studies have shown high rates of acceptability and satisfaction with vaginal ring usage in adult and adolescent women and a high rate of continuation using a traditional start method (6).

The "quick start" method of initiating use of OCs has been found to improve continuation rates and overall method satisfaction compared to traditional start in large studies of adult women (7) and also in small studies of adolescents (8) without significantly affecting incidence of breakthrough bleeding or patient satisfaction (9). "Quick start" contraceptive vaginal ring has been studied in women aged 18-40 years and found to have a more favorable bleeding profile than "quick start" Ortho-Tricyclen Lo (10). This decreased incidence of altered bleeding may be a more favorable benefit of "quick start" contraceptive vaginal ring in the adolescent population as well.

One of the biggest obstacles to use of the contraceptive vaginal ring in clinical practice is having the patient overcome the idea of vaginally inserting the ring, especially in the adolescent population (11). It seems logical that initiating the vaginal ring in the office via the "quick start" method may improve patient acceptance and comfort with the method, thus improving continuation rates in these patients compared to traditional initiation.

We propose to perform a randomized controlled trial comparing "quick start" to traditional start NuvaRing in adolescents. Subjects meeting inclusion criteria will be randomized to either start the method in the office immediately or start the method within 5 days of her next menstrual period. Subjects will follow up at 3, 6, and 12 months, at which time we will assess continuation, bleeding patterns, pregnancy, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria: 1) female aged 15 through 21 presenting for contraception; 2) willing to use the NuvaRing as their contraceptive method; 3) English-speaking; 4) up to date on routine health maintenance screening (pap smear within 3 years of initiation of sexual intercourse and Gonorrhea/ Chlamydia testing yearly or with each new partner); and 5) able to read and understand the consent form.

Exclusion Criteria: 1) are pregnant; 2) have a contraindication to hormonal contraception; 3) are unwilling to use NuvaRing as their contraceptive method; 4) are currently using any hormonal contraceptive or have used one within past 2 months; 5) have used emergency contraception in the past 7 days; 6) have had unprotected intercourse in the past 10 days; 7) have untreated Gonorrhea or Chlamydia; or 8) are unable to give informed consent because of psychiatric or cognitive problems.

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole W Karjane, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Not planned.

REFERENCES:
- [Background] Zibners A, Cromer BA, Hayes J. Comparison of continuation rates for hormonal contraception among adolescents. J Pediatr Adolesc Gynecol. 1999 May;12(2):90-4. doi: 10.1016/s1083-3188(00)86633-4. PMID 10326194
- [Background] Rosenberg M, Waugh MS. Causes and consequences of oral contraceptive noncompliance. Am J Obstet Gynecol. 1999 Feb;180(2 Pt 2):276-9. doi: 10.1016/s0002-9378(99)70718-0. PMID 9988830
- [Background] van den Heuvel MW, van Bragt AJ, Alnabawy AK, Kaptein MC. Comparison of ethinylestradiol pharmacokinetics in three hormonal contraceptive formulations: the vaginal ring, the transdermal patch and an oral contraceptive. Contraception. 2005 Sep;72(3):168-74. doi: 10.1016/j.contraception.2005.03.005. PMID 16102549
- [Background] Rivera R, Cabral de Mello M, Johnson SL, Chandra-Mouli V. Contraception for adolescents: social, clinical and service-delivery considerations. Int J Gynaecol Obstet. 2001 Nov;75(2):149-63. doi: 10.1016/s0020-7292(01)00371-x. PMID 11684110
- [Background] Novak A, de la Loge C, Abetz L, van der Meulen EA. The combined contraceptive vaginal ring, NuvaRing: an international study of user acceptability. Contraception. 2003 Mar;67(3):187-94. doi: 10.1016/s0010-7824(02)00514-0. PMID 12618252
- [Background] Oddsson K, Leifels-Fischer B, de Melo NR, Wiel-Masson D, Benedetto C, Verhoeven CH, Dieben TO. Efficacy and safety of a contraceptive vaginal ring (NuvaRing) compared with a combined oral contraceptive: a 1-year randomized trial. Contraception. 2005 Mar;71(3):176-82. doi: 10.1016/j.contraception.2004.09.001. PMID 15722066
- [Background] Westhoff C, Kerns J, Morroni C, Cushman LF, Tiezzi L, Murphy PA. Quick start: novel oral contraceptive initiation method. Contraception. 2002 Sep;66(3):141-5. doi: 10.1016/s0010-7824(02)00351-7. PMID 12384200
- [Background] Lara-Torre E, Schroeder B. Adolescent compliance and side effects with Quick Start initiation of oral contraceptive pills. Contraception. 2002 Aug;66(2):81-5. doi: 10.1016/s0010-7824(02)00326-8. PMID 12204779
- [Background] Westhoff C, Morroni C, Kerns J, Murphy PA. Bleeding patterns after immediate vs. conventional oral contraceptive initiation: a randomized, controlled trial. Fertil Steril. 2003 Feb;79(2):322-9. doi: 10.1016/s0015-0282(02)04680-0. PMID 12568841
- [Background] Westhoff C, Osborne LM, Schafer JE, Morroni C. Bleeding patterns after immediate initiation of an oral compared with a vaginal hormonal contraceptive. Obstet Gynecol. 2005 Jul;106(1):89-96. doi: 10.1097/01.AOG.0000164483.13326.59. PMID 15994622

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Start: NuvaRing: Initiation of NuvaRing for contraception per package insert
- Quick Start: NuvaRing: Initiation of NuvaRing for contraception on day of enrollment
Period: Overall Study
Arm/Group | Traditional Start | Quick Start
Started | 31 | 17
Completed | 8 | 5
Not Completed | 23 | 12
Not completed — Lost to Follow-up | 23 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Start | Quick Start | Total
Number analyzed (Participants) | 31 | 17 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 26 | 11 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (1.7) | 18 (2.1) | 18 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants] — all female participants
  Participants
    Female | 31 | 17 | 48
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 11 | 29
  White | 11 | 5 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 31 | 17 | 48

OUTCOME MEASURES:

1. Primary Outcome: Continuation With the Contraceptive Method
Description: Participants reporting continuation with contraceptive method at 3 months
Time Frame: 3 months
Population: Number using method at 3 months
Measure: Number; unit: participants
Groups:
- Quick Start: Start method day of enrollment
  NuvaRing: Initiation of NuvaRing for contraception
Arm/Group | Quick Start | Traditional Start
Number analyzed (Participants) | 17 | 31
participants | 5 | 11

2. Primary Outcome: Method Continuation at 6 Months
Description: Participants reporting continuation of method at 6 months
Time Frame: 6 months
Population: Participants enrolled
Measure: Number; unit: participants
Arm/Group | Traditional Start | Quick Start
Number analyzed (Participants) | 31 | 17
participants | 7 | 2

3. Primary Outcome: Method Continuation at 12 Months
Description: Participants reporting continuation with method at 12 months
Time Frame: 12 months
Population: Participants enrolled
Measure: Number; unit: participants
Arm/Group | Quick Start | Traditional Start
Number analyzed (Participants) | 17 | 31
participants | 0 | 2

4. Secondary Outcome: Pregnancy
Description: Number of pregnancies reported
Time Frame: 3,6, and 12 mo
Population: There were no reported pregnancies during the study period
Measure: Number; unit: participants
Arm/Group | Quick Start | Traditional Start
Number analyzed (Participants) | 17 | 31
participants | 0 | 0

5. Secondary Outcome: Bleeding Profile
Time Frame: 3, 6, and 12 months
Population: None of the participants returned their menstrual calendars to assess this outcome
Arm/Group | Quick Start | Traditional Start
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Satisfaction
Description: Rating of patient satisfaction with method
Time Frame: 3, 6, and 12 months
Population: None of the participants returned their satisfaction survey
Arm/Group | Quick Start | Traditional Start
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Traditional Start | Quick Start
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/17
Other Adverse Events (participants affected / at risk) | 0/31 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No